CLINICAL TRIAL: NCT05452096
Title: A Randomized Controlled Trial Investigating the Effects of a Multimodal Shift-work Intervention on Drivers' Fatigue, Sleep, Health and Performance Parameters.
Brief Title: SHIFTPLAN: an RCT Investigating the Effect of a Shift Work Intervention on Fatigue, Sleep and Health.
Acronym: SHIFTPLAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EDGE 000339
Record Dates: First submitted 2022-06-20; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: Shift-work Disorder; Insomnia; Fatigue; Mental Health Issue; Quality of Life; Coping Skills; Circadian Rhythm Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue; Chronobiology Disorders

STUDY DESIGN:
Intervention Model Description: SHIFTPLAN is a randomized controlled interventional trial. It can be situated in occupational health and field research. The drivers will be 1:1 randomized to either the intervention or the control group according to a parallel group design.
Who Masked: Investigator, Outcomes Assessor
Masking Description: After the intake visit with the occupational health physician (OHP) of the relevant service region, all data of the drivers that have agreed to participate and have given their informed consent will be coded, and therefore encrypted data will be sent to the PI for further evaluation.
  The stratified randomization will be done by Qminim a web-based randomization system which uses minimization to ensure a similar distribution of the stratifying factors between the study conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention provided to the intervention group is based on evidence-based good standard of care and includes:
  * Healthy scheduling (fast forward-rotating shift schedules adapted to chronotype, adequate resting times, napping, bright-light therapy)
  * Education program for drivers (psychoeducation promoting sleep hygiene, cognitive-behavioral strategies, stress-management techniques, information on chronotherapy such as bright-light therapy and napping)
  Interventions: Behavioral: Education program and ergonomic schedulling
- Control group (No Intervention): The control group will continue working according to the default shift schedules while being assigned to a waiting list in anticipation of the education program.

INTERVENTIONS:
Behavioral: Education program and ergonomic schedulling — The duration: six months. The explicit choice for a multimodal intervention to be tested as a whole is in line with the assertion of other experts that workplace interventions using a single approach will not be effective.
  Multimodal intervention
  1. Implementing healthy scheduling. This will imply fast forward-rotating shift schedules, being adapted to chronotype, allowing for adequate resting times between shifts and series of shifts, allowing for napping at work, in particular during the first two days of an early shift.
  2. Education program for drivers: psychoeducation on the sleep-wake cycle chronotypes, based on the cognitive-behavioral treatment of insomnia (CBT-i), information on the impact of light on wakefulness and sleep, information on napping and creating awareness on daytime sleepiness, tools for stress reduction, physical exercise, information on healthy eating in the context of shiftwork The education program will consist of a one-day, 8-hour session.
  Arms: Intervention group

SUMMARY:
Shift work is associated with disturbed life rhythms resulting from chronic exposure to circadian misalignment and sleep restriction, with long-term participation in most shift schedules causing serious health problems. Epidemiological data show that shift workers are at increased risk of sleepiness, fatigue and insomnia, cardiovascular disease, breast cancer and shift-work disorder. Prevalence estimates of shift-work disorder vary between 5% and 26,5%.

Given these widespread and serious health and functional consequences of shift work, there is a necessity for treatments that improve shift workers' health and work performance. Most non-pharmacological recommendations mention improved scheduling, bright-light exposure, napping, psychoeducation fostering sleep hygiene, and cognitive-behavioral interventions.

The effects of shift work on the health, fatigue and sleepiness of drivers have been robustly investigated in observational studies, as well as the effects of single measures such as scheduling or resting times. But studies on the effectiveness of countermeasures against the adverse impact of shift work are sparse, especially for high-risk populations such as professional drivers and controlled intervention studies are lacking. Several other investigators expounded the need for a multi-level approach to managing occupational sleep-related fatigue and workplace interventions to promote sleep and health of shift workers. Highlighting the high public-health burden associated with lack of recuperative sleep, the authors pointed out the pressing need to develop policies and implement programs aimed at improving workers' sleep health.

With SHIFTPLAN, the investigators aim to fill this gap in comprehensive approaches. To their knowledge, this is the first randomised controlled trial to systematically gauge the effect of a multimodal program that includes ergonomic shift scheduling and an educational program on well-defined health, sleep and performance outcomes in professional drivers.

DETAILED DESCRIPTION:
The duration of the intervention will be six months. The intervention provided to the intervention group is based on evidence-based good standard of care and includes: 1) Healthy scheduling (fast forward-rotating shift schedules adapted to chronotype, adequate resting times, napping, bright-light therapy); 2) Education program for drivers (psychoeducation promoting sleep hygiene, cognitive-behavioral strategies, stress-management techniques, information on chronotherapy such as bright-light therapy and napping) The control group or "waiting-list group" will include drivers who will continue working according to the default shift schedules while being assigned to a waiting list in anticipation of the education program to which they will able to suscribe after completing the study.

ELIGIBILITY:
Inclusion Criteria:

* - Professional drivers having worked in shifts with the transport company in full-time or ≥80% part-time employment in the company's regular backward-rotating schedule for at least two years.

Exclusion Criteria:

* Regular medication for high blood pressure and uncontrolled high blood pressure (defined as exceeding 140/90 mmHg) at screening, regular medication for diabetes, sleeping pills or sedative medication for depression (defined as trazodone, mirtazapine and amitriptyline). Because our secondary outcomes imply the evolution of blood-pressure and blood-sugar parameters, drivers with such pre-existing controlled or non-controlled comorbidity will not be eligible for participation.
* High risk of moderate-to-severe obstructive sleep apnea syndrome (OSAS) as assessed with the STOP-Bang questionnaire, a simple, easy to remember and self-reportable screening tool. We will use a cut-off score of 6 or higher to indicate the presence of OSAS.
* Drivers combining their job as a professional driver with another job elsewhere.
* Excessive sleepiness as defined as a score in excess of 12 on the Epworth Sleepiness Scale (ESS). Although the habitual cut-off is >9, we opted for this higher threshold because we will be examining the effect of the intervention on daytime sleepiness. All applicants with an ESS >12 will be excluded and referred to a general practitioner for further evaluation.
* A BMI higher than 35. We chose this cut-off value based on the data provided by the external occupational health service, which showed that in 2018, 42.6 % of their drivers had a mean BMI of 25-30 and 27.5 % a BMI between 30-40.
* The presence of major depression as defined by a score exceeding the threshold of 1.75 on the Hopkins Symptom Checklist (HSCL-25), where higher scores were demonstrated to be highly indicative of depressive disorder according to the DSM-5 and characterized as "a case requiring treatment".

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change in sleepiness as assessed with the Epworth Sleepiness Scale (ESS). | Assessed at baseline and monthly up to and including the final 6-month evaluation and the statistical relevance of improvement (first to last score).
  The Epworth Sleepiness Scale (ESS) is a validated self-report scale that gauges daytime sleepiness. The eight items of the ESS ask the respondent how likely (s)he is to doze off or fall asleep in different situations of everyday life. Total scores can range from 0 to 24 and ESS scores exceeding 9 are considered indicative of daytime sleepiness. A drop of 2,5 units will be considered a clinical minimally important difference.

SECONDARY OUTCOMES:
Effect on fatigue indices of the drivers as assessed with the CIS (Checklist Individual Strength). It is to be noted that fatigue and sleepiness are two distinct states of being that may be present or absent independently from each other, whe | Evolution of CIS scores from baseline to three and six months and the statistical relevance of improvement (first to last score).
  The CIS (Checklist Individual Strength) The CIS is a validated, self-administered questionnaire assessing fatigue. It consists of 20 statements for which the respondent has to indicate on a 7-point Likert-scale to what extent the particular statement applies to him or her. The final score is obtained by adding the scores to all questions (range 20-140), where scores of 27 or higher are taken to indicate abnormal fatigue and scores ≥35 severe fatigue. Scores in excess of 76 have been associated with a high risk of chronic absenteeism in a working population. A drop of 10 units will be considered a clinical minimally important difference.
Sleep outcomes as evaluated by Total sleep time (TST) and sleep efficiency (SE) | Evolution at baseline, three and six months of mean total sleep time (TST) and sleep efficiency (SE)
  As derived from self-recorded sleep-wake patterns by keeping a sleep-wake diary
Sleep outcomes measured as scores on the Pittsburgh Sleep Quality Index (PSQI). | scores on the PSQI at baseline, three and six months and the statistical relevance of the baseline to 6-month change
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances. Although self-rated, the PSQI is widely used to assess sleep in sleep and shift-work research, where a global PSQI score >5 is indicative of poor sleep.
General health-related quality of life (HR-QoL) as assessed with the SF-36 | evolution of total SF-36 scores from baseline to three and six months and the statistical relevance of first-to-last score improvement
  The SF-36 The SF-36 is one of the most widely used generic self-report measures of health-related quality of life and consists of 36 items that are structured into nine subscales. The scales are scored from 0-100 (transformed scale = (actual raw score - lowest possible raw score)/possible raw score range) x 100), with higher scores indicating better health.
Absenteeism: sick leave in terms of number of days off work due to illness will be derived from official records of and provided by the company | Data from baseline and after six months
  Absenteeism: formal data collected and provided by the company.
Clinical health outcome: evolution of blood pressure as measured in mmHg | Evolution of blood pressure from baseline, to three and to six months and the statistical relevance of the improvement (first-to-last change).
  Normal blood pressure is defined as a value lower than 140/90 mmHg
Clinical health outcome: evolution of Body Mass Index (BMI) as measured in kg/m² | Evolution of BMI from baseline, to three and to six months and the statistical relevance of the improvement (first-to-last change).
  Normal BMI is defined as a value lower than 25 kg/m²
Clinical health outcome: evolution of fasting blood glucose as measured in mmol/l | Evolution of fasting blood glucose from baseline, to three and to six months and the statistical relevance of the improvement (first-to-last change).
  Normal fasting blood glucose concentration according to the WHO is a value between 3.9 and 5.6 mmol/l
Clinical health outcome: evolution of glycosylated hemoglobin (HbA1c) as measured in mmol/mol | Evolution of HbA1c from baseline, to three and to six months and the statistical relevance of the improvement (first-to-last change).
  On average, normal HbA1c for non-diabetics is < 36 mmol/mol
Clinical health outcome: evolution of high-sensitive C-reactive protein (hsCRP) measured in mg/L | Evolution of hsCRP from baseline, to three and to six months and the statistical relevance of the improvement (first-to-last change).
  High-sensitive C-reactive protein (hsCRP) is shown to be related to cardiovascular health. General guidelines for hsCRP scores: low risk of cardiovascular disease: less than 1.0 mg/L, average risk: 1.0 to 3.0 mg/L, high risk: above 3.0 mg/L
Mood and anxiety as gauged with the Hopkins Symptom Checklist (HSCL-25) | Assessed at baseline and at six months
  This self-administrated questionnaire helps to assess and measure anxiety and depression in multiple settings. Anxiety and depression show considerable overlap in primary-care populations and its brevity and self-report format makes the scale well-suited for use in the busy primary-care setting. The scale's 25 questions are divided into two subsections relating to the presence and intensity of symptoms of depression and anxiety as experienced during the previous week. The final score ranges from 1.00 to 4.00 and is calculated by dividing the sum of the scores of all items by 25. Generally, scores over 1.75 are taken to be indicative of a major depression.

OTHER OUTCOMES:
Correlation between the intervention effects and chronotypes as determined by the Morningness-Eveningness questionnaire (MEQ): Exploratory | 6 months
  This self-assessment scale is used to determine morningness-eveningness in human circadian rhythms and has 19 items subdivided into subscales. MEQ scores are to be added and can vary from 16 to 86. Scores lower or equal to 41 typify respondents as an "evening type", scores exceeding 59 as a "morning type" and scores between 42-58 as a "neutral type"

CONTACTS AND LOCATIONS:
Overall Officials: Filip Van Den Eede, MD, PhD, Study Chair — Antwerp University Hospital (UZA). University of Antwerp (UA); Johan Verbraecken, MD, PhD, Study Chair — Antwerp University Hospital (UZA). University of Antwerp (UA)

REFERENCES:
- [Derived] Declercq I, Van Den Eede F, Roelant E, Verbraecken J. SHIFTPLAN: a randomized controlled trial investigating the effects of a multimodal shift-work intervention on drivers' fatigue, sleep, health, and performance parameters. Trials. 2022 Aug 17;23(1):662. doi: 10.1186/s13063-022-06573-6. PMID 35978435
- Available data/document: Study Protocol: TRLS-D-21-00760R2 — https://trialsjournal.biomedcentral.com/ — Study protocol has been accepted for publication on https://trialsjournal.biomedcentral.com/ . However, BMC requires registration of all clinical trials reported in manuscripts submitted to its journals in a registry listed on the ICMJE website or in any of the primary registries that participate in the WHO International Clinical Trials Registry Platform.